CLINICAL TRIAL: NCT06058533
Title: The Effectiveness of Pre-Visit Positive Imagery in Reducing Dental Anxiety
Brief Title: Pre-Visit Positive Imagery in Reducing Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Catherine Pham, Assistant Professor of Clinical Dentistry, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HS-23-00464
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): No intervention will be given to this group. Each treatment visit will move forward as routine.
- Previsit Imagery Group (Experimental): This group will be given previsit imagery (picture book) before treatment visit.
  Interventions: Other: Previsit Imagery Picturebook

INTERVENTIONS:
Other: Previsit Imagery Picturebook — This picturebook will include pictures of the dental operatory and materials the patient can expect to see during their dental treatment appointment. The pictures included will be generalized pictures of a dental operatory and dental materials. The picture book will also include some words to describe what is happening during the appointment. It is important to note that pictures of the local anesthetic / needle will not be shown in the picture book but will be used during the appointment. The procedures described are standard protocol at both clinics. The traditional picture book shown will be a hard copy.
  Arms: Previsit Imagery Group

SUMMARY:
The purpose of this study is to determine whether pre-visit positive imagery has an impact in decreasing dental anxiety and fear in pediatric patients as well as increasing patient cooperation during treatment visits. Patients needing at least 1 composite filling with nitrous and local anesthetic will receive a picture book if they are selected in the experimental group, and no picture book if they are in the control group. Patients will be asked to be fill out a pre-operative survey and post-operative survey asking how they feel about treatment. Parents will also be asked to fill out a post-operative survey.

DETAILED DESCRIPTION:
This study is a prospective randomized control trial. The study will be conducted at the Herman Ostrow School of Dentistry Pediatric Dental Clinic and Healthy Smiles for Kids of Orange County clinic. Established patients of record that are 4-10 years old who meet the inclusion criteria will qualify.

Participants will be randomly assigned to two groups by flipping a coin and having pre-assigned envelopes in numeric order for each participant. The envelopes will be made ahead of time with heads representing Group 1 and tails representing Group 2. The envelopes will then be numbered and stored in a folder; once a participant consents to enroll in the study, the envelope will be drawn in numeric order determining the participants group number to ensure it is randomized, Group 1 will include patients receiving positive pre-visit imagery. Group 2 will be the control group and will not receive any form of positive pre-visit imagery. The positive pre-visit imagery group 1 will receive a picture book explaining their dental treatment appointment with pictures and some words. The picture book will be a hard copy and will be shown to them by a faculty advisor at USC and by the PI at Healthy Smiles for Kids. The patient's behavior will initially be assessed at their new patient or recall appointment based off the Frankl behavior scale. At the end of the treatment visit, patient behavior will be measured by the dental provider using the Frankl behavior scale. The dentists rating the behavior will be calibrated to ensure there is consistency in the Frankl scale rating and criteria for each score.

Patients will also be asked to fill out a pre- and post-survey that allows them to express their level of dental fear and anxiety before and after the appointment using the Venham Picture Test. The total time commitment will be about 20 minutes and will be a part of their normal dental visit, no additional time is needed. Parents/caregivers will also be given a post-operative survey asking whether they felt the pre-visit positive imagery helped improve patient's behavior.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are healthy with no systemic conditions and are considered ASA I or ASA II
* Patients who have never had any form of dental treatment before.
* Patients who need at least 1 filling to be restored with composite due to caries and will need local anesthetic and nitrous oxide inhalation.
* English speaking patients

Exclusion Criteria:

* Patients with a visual impairment
* Patients with developmental delays that are unable to read or interpret pictures for their age-level.
* Patients whose treatment changes to something other than composite
* Patients who refuse to wear nitrous hood.
* Patients who are unable to read and comprehend English.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Dental Anxiety | 1 day (1 hour during their dental visit)
  Patients will also be asked to fill out a pre- and post-survey that allows them to express their level of dental fear and anxiety before and after the appointment using the Venham Picture Test. The total time commitment will be about 20 minutes and will be a part of their normal dental visit, no additional time is needed.
Patient Behavior | 1 day (1 hour during their dental visit)
  Parents/caregivers will also be given a post-operative survey asking whether they felt the pre-visit positive imagery helped improve patient's behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Arusha Bhatia, Principal Investigator — Herman Ostrow School of Dentistry of USC
Locations (1):
- Herman Ostrow School of Dentistry of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No